CLINICAL TRIAL: NCT02911662
Title: Treatment of Asymptomatic Bacteriuria in Pregnancy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to enroll patients at anticipated rate.
Sponsor: Trinity Health Michigan (Other)
Responsible Party: Principal Investigator, Pooja Green, Director of Obstetrical Research, Trinity Health Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR-16-1661
Record Dates: First submitted 2016-09-15; First posted 2016-09-22 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Bacteriuria (Asymptomatic) in Pregnancy
MeSH Terms: conditions — Bacteriuria | interventions — Cephalexin; Nitrofurantoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3-day treatment (Experimental): Three-day treatment with Cephalexin or Nitrofurantoin for diagnosis of asymptomatic bacteriuria in pregnancy.
  Interventions: Drug: Cephalexin; Drug: Nitrofurantoin
- 7-day treatment (Active Comparator): Seven-day treatment with Cephalexin or Nitrofurantoin for diagnosis of asymptomatic bacteriuria in pregnancy.
  Interventions: Drug: Cephalexin; Drug: Nitrofurantoin

INTERVENTIONS:
Drug: Cephalexin — Cephalexin will be prescribed for women with a positive urine culture but no symptoms of urinary tract infection.
  Other Names: Keflex
Drug: Nitrofurantoin — Macrobid will be prescribed for women allergic to penicillin with a positive urine culture but no symptoms of urinary tract infection.
  Other Names: Macrobid

SUMMARY:
This is a prospective randomized controlled day comparing the efficacy of three-day antimicrobial treatment of asymptomatic bacteriuria (ASB) in pregnancy to the standard seven-day treatment. Half the patients will receive 3-day treatment and the other half will receive 7 days of antibiotics.

DETAILED DESCRIPTION:
The current standard of practice is to treat pregnant patients with ASB with a 7-day course of oral antimicrobial agents. If bacteriuria persists women are retreated with the same of different agent for a second course of 7 to 14 days and they may be subsequently placed on prophylaxis.

In nonpregnant women, an uncomplicated lower urinary tract infection may be treated with a short course regimen from 1 to 3 days. This approach has similar rates of persistent bacteriuria or symptoms following treatment when compared to women treated with a more conventional approach. If the infection recurs or persists, the patient may then be treated with the more traditional 7 to 14 day course. The advantages of single-dose regimens are cost and patient compliance, but a major disadvantage is the failure to eradicate uropathogens from the vaginal reservoir, which results in more frequent early recurrences.

The three-day regimen is advocated to maintain the advantages of lower costs and patient compliance but improving cure rates. Multiple studies have shown the advantage of even a short course of antibiotics as opposed to no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ≥ 18 years of age seeking prenatal care at the Academic Obstetrics and Gynecology Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
* Randomization will occur if the patient every has a urine culture demonstrating ≥10,000 cfu/ml of a pathogenic urinary tract organism

Exclusion Criteria:

* Symptomatic bacteriuria (cystitis or pyelonephritis) at the time of urine collection
* Previously treated bacteriuria in current pregnancy
* Past medical history of known congenital or acquired urinary tract anomaly or abnormality (i.e. pelvic kidney, single kidney, renal transplant)
* Any antibiotic use within the week prior to urine sampling
* Urine culture revealing growth of the following organisms: Lactobacillus, coagulase-negative staphylococcus

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-09; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Evidence that 3-day treatment is as effective as 7-day treatment of asymptomatic bacteriuria in pregnancy. | Within 21 days of treatment
  Comparison of percentage of women in each group with successful treatment or asymptomatic bacteriuria with negative urine culture 2 weeks after randomized treatment.

SECONDARY OUTCOMES:
Comparison of development of cystitis during pregnancy. | Until 6 weeks postpartum
  Comparison of percentage of women in each group who develop cystitis during pregnancy and the postpartum period.
The occurence of preterm delivery | Assessed at the time of delivery
  Comparison of the percentage of women in each group who deliver at <37 weeks gestation.
Comparison of development of pyelonephritis during pregnancy | Until 6 weeks postpartum
  Comparison of percentage of women in each group who develop pyelonephritis during pregnancy and the postpartum period.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph Mercy Hospital, Ypsilanti, Michigan, United States

REFERENCES:
- [Background] Widmer M, Lopez I, Gulmezoglu AM, Mignini L, Roganti A. Duration of treatment for asymptomatic bacteriuria during pregnancy. Cochrane Database Syst Rev. 2015 Nov 11;2015(11):CD000491. doi: 10.1002/14651858.CD000491.pub3. PMID 26560337
- [Background] Patterson TF, Andriole VT. Detection, significance, and therapy of bacteriuria in pregnancy. Update in the managed health care era. Infect Dis Clin North Am. 1997 Sep;11(3):593-608. doi: 10.1016/s0891-5520(05)70375-5. PMID 9378925
- [Background] Romero R, Oyarzun E, Mazor M, Sirtori M, Hobbins JC, Bracken M. Meta-analysis of the relationship between asymptomatic bacteriuria and preterm delivery/low birth weight. Obstet Gynecol. 1989 Apr;73(4):576-82. PMID 2927852